CLINICAL TRIAL: NCT03528967
Title: Enoxaparine en PREvention Des insuffiSAnces Placentaires Chez Les Femmes eNCEintes
Brief Title: Enoxaparin in the Prevention of Placental Insufficiency in Pregnant Women
Acronym: PRESANCE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Les Laboratoires des Médicaments Stériles (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EG01
Record Dates: First submitted 2018-05-07; First posted 2018-05-18 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2018-08

CONDITIONS: Placental Insufficiency; Enoxaparin
MeSH Terms: conditions — Placental Insufficiency | interventions — Enoxaparin; Aspirin; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Patients going on ASPIRIN 100 mg/day combined with ENOXAPARIN 4000 IU per dat prevention treatment according to randomization:
  * Administer Aspirin 100 mg Oral Tablet, Enteric Coated once daily
  * Administer the Enoxaparin preventive dose of 4000 IU as a subcutaneous Enoxaparin 40 mg / 0.4 mL Prefilled Syringe once daily
  * Start treatment from inclusion visit
  * Maintain treatment until the day of delivery, or the appearance of a complication (Retroplacental hematoma (RPH), preeclampsia (PE) , In utero fetal death (IUFD), or Intrauterine growth restriction (IUGR) and its complications)
  Interventions: Drug: Enoxaparin 40 mg / 0.4 mL Prefilled Syringe; Drug: Aspirin 100 mg Oral Tablet, Enteric Coated
- Arm 2 (Other): Patients going on ASPIRIN 100 mg/day prevention treatment alone according to randomization:
  * Administer only Aspirin 100 mg Oral Tablet, Enteric Coated once daily
  * Administer orally
  * Start treatment from inclusion visit
  * Maintain treatment until 35 Weeks of Amenorrhea (WA)
  Interventions: Drug: Aspirin 100 mg Oral Tablet, Enteric Coated

INTERVENTIONS:
Drug: Enoxaparin 40 mg / 0.4 mL Prefilled Syringe
  Arms: Arm 1
Drug: Aspirin 100 mg Oral Tablet, Enteric Coated

SUMMARY:
Assessment of the effectiveness of Enoxaparin, at a preventive dose, combined with Aspirin treatment versus Aspirin only treatment in reducing placental insufficiency in pregnant women.

DETAILED DESCRIPTION:
Randomized, prospective, monocentric, open-label comparative study with two parallel groups (Enoxaparin, at a preventive dose, combined with Aspirin versus Aspirin alone), with the main objective being to evaluate the effectiveness of enoxaparin, at a preventive dose, in reducing placental insufficiency during pregnancy in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and
* Age ≤ 45 years and
* Single and confirmed pregnancy and
* Intrauterine growth restriction (IUGR) history with an estimated fetal weight (ESW) < 3rd percentile and / or
* In utero fetal death (IUFD) history > 12 weeks of amenorrhea (WA) and / or
* Central Retroplacental hematoma (RPH) history < 34 WA and / or
* History of severe preeclampsia < 34 WA and
* Informed consent, written and obtained

Exclusion Criteria:

* Age <18 years or
* Age > 45 years or
* Multiple pregnancy or
* Pregnancy > 7 WA or
* Positive immunological assessment or
* Known history of Thromboembolic diseases, Hemorrhagic diseases, Systemic Lupus Erythematosus (SLE), Heparin-induced thrombocythemia (HIT), Suspicion of thrombophilia (burdened history) or an episode of Deep Vein Thrombosis (DVT) or
* Anticoagulation required or
* Thrombocythaemia < 100,000 plq / µl or
* Weight > 100 kg or
* Osteoporosis or
* Known allergy to the study products or
* Inability to ensure injections' administration or
* Family history of DVT before 40 years of age or

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2013-10-23 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of maternal death | 7 - 42 weeks of amenorrhea
  To compare the incidence of maternal death between the two arms of the study.
Recurrence rate of preeclampsia | 7 - 42 weeks of amenorrhea
  To compare the recurrence rate of preeclampsia between the two arms of the study.
Incidence of intrauterine growth restriction (IUGR) | 7 - 42 weeks of amenorrhea
  To compare the incidence of IUGR between the two arms of the study.
Incidence of retroplacental hematoma (RPH) | 7 - 42 weeks of amenorrhea
  To compare the incidence of RPH between the two arms of the study.
Incidence of perinatal death | 7 - 42 weeks of amenorrhea
  To compare the incidence of perinatal death between the two arms of the study.

SECONDARY OUTCOMES:
Incidence of miscarriage | 13 - 21 weeks of amenorrhea
  To compare the incidence of miscarriage between the two arms of the study.
Incidence of in utero fetal death (IUFD) | 22 weeks of amenorrhea at birth
  To compare the incidence of IUFD between the two arms of the study.
Incidence of neonatal death | From birth to 28 days of life
  To compare the incidence of neonatal death between the two arms of the study.
Number of adverse events | 7 - 42 weeks of amenorrhea
  To compare the safety of both study products

CONTACTS AND LOCATIONS:
Overall Officials: Dalenda Chelly, OB/GYN, Principal Investigator — Wassila Bourguiba Hospital Tunis
Locations (1):
- Maternity Center of Wassila Bourguiba Hospital - Department A, Tunis, Tunisia